CLINICAL TRIAL: NCT02072512
Title: The Study of Goserelin Plus Fulvestrant Comparing With Goserelin Plus Anastrozole for Advanced Breast Cancer
Acronym: PROOF
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Hospital Affiliated to Military Medical Science, Beijing (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 307BC ET-01
Record Dates: First submitted 2014-02-07; First posted 2014-02-26 (Estimated); Last update posted 2014-02-26 (Estimated); Status verified 2014-02

CONDITIONS: Metastatic Breast Cancer
Keywords: pre- and perimenopausal HR+ advanced breast cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — Fulvestrant; Goserelin; Anastrozole

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Fulvestrant (Active Comparator): Goserelin plus High Dose Fulvestrant
  Interventions: Drug: Fulvestrant; Drug: Goserelin
- Anastrozole (Active Comparator): Goserelin plus Anastrozole
  Interventions: Drug: Anastrozole; Drug: Goserelin

INTERVENTIONS:
Drug: Fulvestrant — Fulvestrant 500mg I.M. Once/28days,until progression or unacceptable toxicity develops
  Arms: Fulvestrant
Drug: Goserelin — goserelin 3.6mg subcutaneously every 28(± 3) days
  Arms: Fulvestrant
Drug: Anastrozole — Anastrozole 1mg P.O. once daily, until progression or unacceptable toxicity develops
  Arms: Anastrozole
Drug: Goserelin — goserelin 3.6mg subcutaneously every 28(± 3) days
  Arms: Anastrozole

SUMMARY:
The purpose of this study is to assess the efficacy of goserelin plus fulvestrant 500mg comparing with goserelin plus anastrozole as first line endocrine therapy for pre- and perimenopausal HR+ advanced breast cancer.

DETAILED DESCRIPTION:
Premenopausal advanced breast cancer patients who failed tamoxifen treatment are possible good candidates for ovarian ablation/suppression and aromatase inhibitors.Fulvestrant has been studied little in premenopausal women despite of its attractive mechanism of actions. Based on this rationale, we introduced high-dose of fulvestrant with LHRH agonist as a randomized trial comparing with AI plus LHRH agonist.

To assess efficacy of goserelin plus fulvestrant 500mg comparing with goserelin plus anastrozole as first line endocrine therapy for pre- and perimenopausal HR+ advanced breast cancer in terms of progression-free survival(PFS)

ELIGIBILITY:
Inclusion Criteria:

1. Signed informed consent document on file.
2. All patients must be female with age>18 and premenopausal or perimenopausal.
3. Patients must have an ECOG performance status of 0, 1, or 2.
4. Patients with life expectancy of more than 3 months.
5. Patients with metastatic or locally advanced disease not amenable to therapy with curative intent.
6. Histological/cytological confirmation of breast cancer. Patients must have either positive estrogen and/or progesterone receptor determination by IHC or competitive binding assay on advanced disease, or if not performed on their advanced disease a positive result on their primary breast cancer specimen (Positivity is defined as an Allred score from 3 to 8 by IHC or at least 1% positive tumor nuclei in the sample in the presence of expected reactivity of internal and external controls [35]).
7. Patients who recurred on or after completion of adjuvant tamoxifen therapy(with or without GnRHa). Toremifene could be substituted for tamoxifen in adjuvant setting.
8. Duration of adjuvant tamoxifen(toremifene) treatment should be at least 48 weeks or more.
9. Patients with measurable lesion at baseline, or Patients with bone lesions, lytic or mixed (lytic + sclerotic), in the absence of measurable disease as defined by RECIST 1.1 criteria
10. Patients may receive irradiation to any bony sites of disease for pain control or for prevention of fracture.
11. For women of childbearing potential, agreement to use one highly effective form of non-hormonal contraception or two effective forms of non-hormonal contraception by the patient and/or partner and to continue its use for the duration of study treatment and for 6 months after the last dose of study treatment.

Exclusion Criteria:

1. Presence of life-threatening metastatic visceral disease, defined as extensive hepatic involvement, or any degree of brain or leptomeningeal involvement (past or present), or symptomatic pulmonary lymphangitic spread. Patients with discrete pulmonary parenchymal metastases are eligible, provided their respiratory function is not compromised as a result of disease.
2. Postmenopausal woman, defined as a woman fulfilling any 1 of the following criteria:

   * Age .60 years
   * Prior bilateral oophorectomy
   * Age<60 years and amenorrheic for 12 or more months in the absence of chemotherapy, tamoxifen, toremifene, or ovarian suppression and FSH and estradiol in the postmenopausal range(according to local sites).
   * If taking tamoxifen or toremifene, and age<60 years, then FSH and plasma estradiol level in postmenopausal ranges(according to local sites).
3. More than one regimen of chemotherapy for advanced disease.
4. Previous endocrine therapy for advanced disease.
5. Prior treatment with an aromatase inhibitor or fulvestrant.
6. Prior treatment with a GnRHa within 3 months.
7. Treatment with a non-approved or experimental drug within 4 weeks before randomisation.
8. Current or prior malignancy within previous 3 years (other than breast cancer or adequately treated basal cell or squamous cell carcinoma of the skin or in-situ carcinoma of the cervix).
9. History of bleeding diathesis (i.e., disseminated intravascular coagulation [DIC], clotting factor deficiency), or long-term anticoagulant therapy.
10. Known hypersensitivity to the active substance or to any of the excipients of this product, or other GnRHa.
11. HER-2 over-expressing breast cancer and concomitant trastuzumab treatment.
12. Pregnancy and lactation.
13. Any severe concomitant condition which makes it undesirable for the patient to participate in t he trial or which would jeopardize compliance with the trial protocol. e.g., uncontrolled cardiac disease, uncontrolled diabetes mellitus, severe osteoporosis or renal failure and so on .
14. Inadequate organ function

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 180 (Estimated)
Dates: Start 2014-01; Primary Completion 2015-11 (Estimated); Study Completion 2016-12 (Estimated)

PRIMARY OUTCOMES:
the efficacy of goserelin plus fulvestrant 500mg and the efficacy of goserelin plus anastrozole as first line endocrine therapy for pre- and perimenopausal HR+ advanced breast cancer in terms of progression-free survival(PFS) | Progression-free survival (PFS) is defined as the time elapsed between randomization and tumor progression(by RECIST version 1.1) or death from any cause.Participants will be followed for an expected average of 1 year.
  Primary endpoint is progression-free survival. Progression-free survival (PFS) is defined as the time elapsed between randomization and tumor progression(by RECIST version 1.1) or death from any cause

SECONDARY OUTCOMES:
the overall response rate(by RECIST version 1.1) of patients treated with goserelin plus fulvestrant 500mg and the overall response rate of patients treated with goserelin plus anastrozole. | Participants will be followed for an expected average of 1 year.
  to compare overall response rate of patients treated with goserelin plus fulvestrant 500mg with overall response rate of patients treated with goserelin plus anastrozole.
the clinical benefit rate of patients treated with goserelin plus fulvestrant 500mg and clinical benefit rate of patients treated with goserelin plus anastrozole. | Participants will be followed for an expected average of 1 year.

OTHER OUTCOMES:
the duration of response of patients treated with goserelin plus fulvestrant 500mg and duration of response of patients treated with goserelin plus anastrozole. | Participants will be followed for an expected average of 1 year.
the duration of clinical benefit of patients treated with goserelin plus fulvestrant 500mg and duration of clinical benefit of patients treated with goserelin plus anastrozole. | Participants will be followed for an expected average of 1 year.
the safety and tolerability(by NCI CTCAE v4.0) of goserelin plus fulvestrant 500mg compared with goserelin plus anastrozole. | Participants will be followed for an expected average of 1 year.

CONTACTS AND LOCATIONS:
Overall Officials: Zefei Jiang, Ph.D, Principal Investigator — 307 Hospital of PLA
Locations (1):
- 307 Hospital, Beijing, Beijing Municipality, China